CLINICAL TRIAL: NCT05119621
Title: The Effect of TENS Application Applied Before Mobilization on Pain in Children With Abdominal Surgery: A Randomized Controlled Trial
Brief Title: The Effect of TENS Application for Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUh01a
Record Dates: First submitted 2021-09-03; First posted 2021-11-15 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2022-10

CONDITIONS: Appendicitis Surgery; Inguinal Surgery
Keywords: Transcutaneous Electric Nerve Stimulation; Child; Surgery; Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS application (Experimental): TENS application will be applied to the experimental group before mobilization after abdominal surgery. TENS will be applied for an average of 40 minutes.
  Interventions: Device: TENS application
- Standard pain management (No Intervention): The control group will receive standard pain treatment without any intervention. The group will not receive any other intervention.

INTERVENTIONS:
Device: TENS application — Assigned Interventions: In addition to the standard pain management applied in the clinic, TENS will be applied to children who have had surgery.
  Other Names: Transcutaneous Electrical Nerve Stimulation
  Arms: TENS application

SUMMARY:
The aim of the study which was planned in a randomized controlled experimental design, it was aimed to determine the effect of Transcutaneous Electrical Nerve Stimulation (TENS) application on pain level before mobilization in the postoperative period in children.

DETAILED DESCRIPTION:
Children can often experience chronic muscle, bone, joint pain, headache and abdominal pain, and acutely experience pain due to postoperative and procedural procedures. Effective management of childhood pain is emphasized as a health priority by the World Health Organization and pain communities. The findings of various epidemiological studies emphasized that a significant proportion (49% to 64%) of children receiving treatment in a hospital setting received inadequate pain management services despite the increase in available knowledge and treatments. One of the situations in which pediatric patients encounter acute pain is the postoperative period. Mobilization is delayed in patients who cannot provide adequate pain control, and accordingly, serious complications such as impaired tissue perfusion, atelectasis and deep vein thrombosis may develop. There are studies on the use of TENS, one of the methods used in non-pharmacological pain management, in postoperative pain management in adults. Studies on pain management in children for TENS application are very limited today. There was no evidence for the effectiveness of TENS application applied before mobilization in the postoperative period in children.

ELIGIBILITY:
Inclusion Criteria:

* Be in the 7-12 age range
* Abdominal surgery indication (appendicitis or inguinal region surgery)
* Volunteering to participate in the study
* Receiving monotherapy treatment for epilepsy
* To be able to communicate in Turkish

Exclusion Criteria:

* Administering analgesic therapy other than routine administration
* Patients who have difficulties in mobilization/complications during the operation will be excluded from the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Child Introduction Form | (First measurement-After the operation, when the patient is taken to her bed and fully awakened)
  The introductory information form was prepared by the researcher in line with the literature information. The introductory information form consists of 10 questions covering the characteristics of children and their families (age, gender, parental age, education level, family type, income status), and operational characteristics (patient's complaints, type of surgery, previous operation experience).
Children's Fear Scale | (First measurement-40 minutes on average before mobilization)
  The mean score of the scale, which was translated into Turkish by five independent linguists, was 1.9 ± 0.1 (min=0, max=4). The scale can also be scored by the parent and the researcher. The scale consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety).
Children's Fear Scale | (Second measurement-1 minute on average before mobilization)
  The mean score of the scale, which was translated into Turkish by five independent linguists, was 1.9 ± 0.1 (min=0, max=4). The scale can also be scored by the parent and the researcher. The scale consists of five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety).
Visual Analogue Scale | (First measurement-40 minutes on average before mobilization)
  The scale consists of a horizontal or vertical ruler, 10 cm or 100 mm in length, showing "painlessness" at one end and "the most severe pain" at the other end. For children over the age of six, this scale is reported to be an easy-to-understand and easy-to-apply scale.
Visual Analogue Scale | (Second measurement-1 minute on average before mobilization)
  The scale consists of a horizontal or vertical ruler, 10 cm or 100 mm in length, showing "painlessness" at one end and "the most severe pain" at the other end. For children over the age of six, this scale is reported to be an easy-to-understand and easy-to-apply scale.
The Wong-Baker Faces Pain Rating Scale | (First measurement-40 minutes on average before mobilization)
  In this scale, there are six facial expressions representing the increasing pain intensity from 0 to 5 from left to right. Six facial expressions are scored between 0-5 points from left to right (0 points = very happy/no pain, 5 points = indicates the most severe pain). As the score obtained from the scale increases, pain tolerance decreases, and as the score decreases, the tolerance increases.
The Wong-Baker Faces Pain Rating Scale | (Second measurement-1 minute on average before mobilization)
  In this scale, there are six facial expressions representing the increasing pain intensity from 0 to 5 from left to right. Six facial expressions are scored between 0-5 points from left to right (0 points = very happy/no pain, 5 points = indicates the most severe pain). As the score obtained from the scale increases, pain tolerance decreases, and as the score decreases, the tolerance increases.

CONTACTS AND LOCATIONS:
Overall Officials: Metin GUNDUZ, Md., Study Director — Selcuk University; Sibel KUCUKOGLU, PhD., Study Chair — Selcuk University; Hilal KURT SEZER, Lecturer, Principal Investigator — KTO Karatay University; Bayram Sonmez UNUVAR, Principal Investigator — KTO Karatay University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Ali S, Chambers A, Johnson DW, Newton AS, Vandermeer B, Williamson J, Curtis SJ. Reported practice variation in pediatric pain management: a survey of Canadian pediatric emergency physicians. CJEM. 2014 Sep;16(5):352-60. doi: 10.2310/8000.2013.131261. PMID 25227643
- [Background] Curtis S, Wingert A, Ali S. The Cochrane library and procedural pain in children: an overview of reviews. Evid Based Child Health. 2012;7(5):1363-99.
- [Background] Elboim-Gabyzon M, Andrawus Najjar S, Shtarker H. Effects of transcutaneous electrical nerve stimulation (TENS) on acute postoperative pain intensity and mobility after hip fracture: A double-blinded, randomized trial. Clin Interv Aging. 2019 Oct 29;14:1841-1850. doi: 10.2147/CIA.S203658. eCollection 2019. PMID 31754300
- [Background] Engen DJ, Carns PE, Allen MS, Bauer BA, Loehrer LL, Cha SS, Chartrand CM, Eggler EJ, Cutshall SM, Wahner-Roedler DL. Evaluating efficacy and feasibility of transcutaneous electrical nerve stimulation for postoperative pain after video-assisted thoracoscopic surgery: A randomized pilot trial. Complement Ther Clin Pract. 2016 May;23:141-8. doi: 10.1016/j.ctcp.2015.04.002. Epub 2015 Apr 20. PMID 25935320
- [Background] Fiorelli A, Morgillo F, Milione R, Pace MC, Passavanti MB, Laperuta P, Aurilio C, Santini M. Control of post-thoracotomy pain by transcutaneous electrical nerve stimulation: effect on serum cytokine levels, visual analogue scale, pulmonary function and medication. Eur J Cardiothorac Surg. 2012 Apr;41(4):861-8; discussion 868. doi: 10.1093/ejcts/ezr108. Epub 2011 Dec 16. PMID 22219414
- [Background] Gerçeker GÖ, Ayar D, Özdemir Z, Bektaş M. Çocuk Anksiyete Skalası-Durumluluk ve Çocuk Korku Ölçeğinin Türk Diline Kazandırılması DEUHFED 2018, 11 (1), 9-13
- [Background] Karakoç S. Açık Kalp Cerrahisi Sonrası Klasik Metodlarla Ağrı Kontrolünün, Alternatif (TENS) Yöntemle Karşılaştırılarak, Hemşire Takip ve Kontrolün Katkısının Araştırılması. Afyon Kocatepe Üniversitesi Sağlık Bilimleri Fakültesi, Yüksek Lisans Tezi, 2009.
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Tokuda M, Tabira K, Masuda T, Nishiwada T, Shomoto K. Effect of modulated-frequency and modulated-intensity transcutaneous electrical nerve stimulation after abdominal surgery: a randomized controlled trial. Clin J Pain. 2014 Jul;30(7):565-70. doi: 10.1097/AJP.0b013e31829ea151. PMID 24901753
- See also: American Academy of Pediatrics, Pain Management in Infants, Children, Adolescents and Individuals with Special Health Care Needs, 2018, — https://www.aapd.org/media/Policies_Guidelines/BP_Pain.pdf